CLINICAL TRIAL: NCT05485662
Title: Remineralization of Molar Incisor Hypomineralization (MIH) With a Hydroxyapatite Toothpaste - an in Situ Study
Brief Title: Remineralization of Molar Incisor Hypomineralization (MIH) With a Hydroxyapatite Toothpaste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Dr. Kurt Wolff GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HSC20210570H
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Remineralization; Hydroxyapatite; Sodium fluoride
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, sequential, single center, controlled clinical trial.
Who Masked: Participant, Investigator
Masking Description: The study will be blinded to both the study team and the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MIH-bearing tooth block exposed to HAP toothpaste (Other): A block of molar incisor hypomineralization (MIH) is mounted in an oral appliance and fitted in the subject for testing with the HAP toothpaste
  Interventions: Other: Hydroxyapatite toothpaste
- MIH-bearing block exposed to Sodium Fluoride toothpaste (Other): A block of molar incisor hypomineralization (MIH) is mounted in an oral appliance and fitted in the subject for testing with the sodium fluoride toothpaste
  Interventions: Other: Sodium Fluoride Toothpaste

INTERVENTIONS:
Other: Hydroxyapatite toothpaste — 10% Hydroxyapatite toothpaste
  Other Names: HAP toothpaste
  Arms: MIH-bearing tooth block exposed to HAP toothpaste
Other: Sodium Fluoride Toothpaste — 1450 parts per million sodium fluoride toothpaste
  Other Names: NaF toothpaste
  Arms: MIH-bearing block exposed to Sodium Fluoride toothpaste

SUMMARY:
This study tests the remineralization of donor teeth (donorMIH) in situ in participants using 10% hydroxyapatite (HAP) toothpaste and sodium fluoride toothpaste.

DETAILED DESCRIPTION:
Prior to each 2-week treatment phase, subjects will complete a 1-week washout period. Following the washout period, the intra-oral appliance containing a donorMIH tooth block will be fitted to each subject by a qualified dentist. Immediately after fitting of the first appliance (on day 1 of the first treatment phase), each subject will receive a soft bristled manual toothbrush for use throughout the duration of the study and a toothpaste according to the treatment phase. Subjects will be instructed to brush their teeth with the appliance in the mouth, two times daily, for 3 minutes on each brushing episode, in the morning after breakfast and last thing before bed, then rinsing with 10 ml of water. Over the study period, all subjects will maintain their normal dietary habits.

A 7-day washout period without an appliance will follow. After completion of the second washout period, subjects will return to the clinic, and the appliance, with another MIH-bearing tooth blocks mounted, will be fitted to the subject for the phase 2 treatment period. This procedure will then be repeated until the 2-week treatment phase is completed, and each subject has gone through the two arms of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* Good general health
* No known history of allergy to personal care/consumer products
* Minimum of 20 natural uncrowned teeth (excluding third molars)
* Normal salivary flow rate (stimulated and unstimulated flow of ≥0.7 ml/min and ≥0.2 ml/min respectively
* Able to consent
* Availability throughout entire study
* Willing to wear intra-oral appliance 24 hours per day
* Willing to use only assigned products for oral hygiene for duration of study

Exclusion Criteria:

* Advanced periodontal disease
* A medical condition that requires pre-medication prior to dental visits/procedures
* Impaired salivary function
* Orthodontic retainer(s)
* Too few teeth to secure the oral appliance
* Disease of the soft or hard oral tissues
* Use of drugs that can affect salivary flow
* Use of antibiotics one month prior to or during this study
* Participation in another clinical study one week prior to the start of washout period or during this study period
* Allergic hisotry to common toothpaste ingredients
* Compromised immune system (HIV, AIDS, Immunosuppressive drug therapy)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bennett T Amaechi, BDS, MS, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- School of Dentistry, University of Texas Health Science Center, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were consented and assessed for eligibility prior to inclusion into the study, and included adults over 18 years of age. Subjects were originally assigned to one of the toothpastes, then after using that toothpaste for 2 weeks, they were assigned to the other toothpaste.
Groups:
- MIH-bearing Tooth Block Exposed to HAP Toothpaste Then Sodium Fluoride Toothpaste: A block of molar incisor hypomineralization (MIH) is mounted in an oral appliance and fitted in the subject for testing with the HAP toothpaste followed by a washout period and then the sodium fluoride toothpaste.
- MIH-bearing Block Exposed to Sodium Fluoride Toothpaste Then the HAP Toothpaste: A block of molar incisor hypomineralization (MIH) is mounted in an oral appliance and fitted in the subject for testing with the sodium fluoride toothpaste then after a washout period, to the HAP toothpaste
Period: Phase 1 Allocation
Arm/Group | MIH-bearing Tooth Block Exposed to HAP Toothpaste Then Sodium Fluoride Toothpaste | MIH-bearing Block Exposed to Sodium Fluoride Toothpaste Then the HAP Toothpaste
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | MIH-bearing Tooth Block Exposed to HAP Toothpaste Then Sodium Fluoride Toothpaste | MIH-bearing Block Exposed to Sodium Fluoride Toothpaste Then the HAP Toothpaste
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Phase 2 Allocation
Arm/Group | MIH-bearing Tooth Block Exposed to HAP Toothpaste Then Sodium Fluoride Toothpaste | MIH-bearing Block Exposed to Sodium Fluoride Toothpaste Then the HAP Toothpaste
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Enrollment: A block of molar incisor hypomineralization (MIH) is mounted in an oral appliance and fitted in the subject for testing with the HAP toothpaste. Subjects are randomized to either hydroxyapatite toothpaste (10%) or sodium flouride (1450 parts per million) toothpaste
Arm/Group | Overall Study Enrollment
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 50.2 [25 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Mineral Density (MD) of Tooth
Description: Images will be collected from the samples to measure the mineral density before and after remineralization treatment. Total number of subjects enrolled in either the first allocation or the second allocation after the washout are included.
Time Frame: Baseline to 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of remineralization
Arm/Group | MIH-bearing Tooth Block Exposed to HAP Toothpaste | MIH-bearing Block Exposed to Sodium Fluoride Toothpaste
Number analyzed (Participants) | 15 | 15
percentage of remineralization
  Combined data | 26.02 (20.68) | 14.64 (9.60)
  Etched | 29.26 (22.99) | 16.83 (9.97)
  Unetched | 16.62 (5.74) | 10.62 (8.13)

ADVERSE EVENTS:
Time Frame: From baseline to study end at 2 weeks
Arm/Group | MIH-bearing Tooth Block Exposed to HAP Toothpaste | MIH-bearing Block Exposed to Sodium Fluoride Toothpaste
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MIH-bearing Tooth Block Exposed to HAP Toothpaste (N=8) | MIH-bearing Block Exposed to Sodium Fluoride Toothpaste (N=7)
Burning (Gastrointestinal disorders) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT05485662/Prot_SAP_000.pdf